CLINICAL TRIAL: NCT03781856
Title: La Vida Buena (The Good Life) Evaluation: A Quasi Experimental Intervention of a Community Health Worker Led Family-based Childhood Obesity Program for Hispanic Children 5-8 Years of Age on the US-Mexico Border
Brief Title: La Vida Buena Childhood Obesity Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Mariposa Community Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1710977008
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Childhood Obesity
Keywords: childhood obesity; intervention; community health workers; community-based
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- La Vida Buena Program (Experimental): Administered in a group setting over the course of 8 weeks in a community setting.
  Interventions: Behavioral: La Vida Buena Program
- Brief educational session (Active Comparator): Administered one on one or in a group setting in a one-hour session at the clinic
  Interventions: Behavioral: Brief Educational Session

INTERVENTIONS:
Behavioral: La Vida Buena Program — The intervention is series of interactive one hour weekly classes over the course of 8 weeks related to child healthy weight, exercise and nutrition. Facilitated by community health workers, the classes are interactive and play-based and designed to engage both the child and accompanying parent or guardian in activities.
  Arms: La Vida Buena Program
Behavioral: Brief Educational Session — A one hour session about nutrition and physical activity to address obesity facilitated by a community health worker
  Arms: Brief educational session

SUMMARY:
Mariposa Community Health Center, a health center in Nogales, Arizona on the US-Mexico border, will provide a program to prevent obesity in children and create a community environment that supports a healthy lifestyle. Mariposa designed and implemented the La Vida Buena ("The Good Life") program and already know that helps families eat more healthily and exercise. Mariposa Community Health Center will test this program on younger children aged 5-8 years old. Providers will refer children who are overweight or obese to the La Vida Buena Program. In order to determine if the La Vida Buena program works, Mariposa Community Health center will implement the 8-week program with 100 overweight or obese children in their Nogales clinic. They will measure their weight (BMI), exercise levels and food habits at the beginning of the program and then 3- months and 6-months after the program ends. Mariposa will compare these results to children in the nearby Rio Rico clinic who do not receive the La Vida Buena program. These 100 overweight or obese children in Rio Rico will instead receive one educational session, and the same information will be collected regarding BMI, exercise level and food habits. After the 6-month period, the children from Rio Rico will be able to receive the full La Vida Buena program.

DETAILED DESCRIPTION:
La Vida Buena is a Mariposa project to educate children and families about healthy eating and exercise habits. The Health providers at Mariposa Nogales and Rio Rico clinics will refer children between 5-8 years old who are overweight or obese and their parents. Each child must participate with a parent or adult caregiver who is at least 18 years old. Before the program begins, the participant will attend an informational consent/registration session where they will be asked to sign a consent form for themselves and their child if they want to participate. The study will ask for certain information from each participant in order to determine if the program is working. Each family will respond to a questionnaire at three points: at the beginning of the program, three months after beginning the program, and six months after beginning the program, for a total of six months.

The questionnaire will include questions about fruit, vegetable and carbohydrate consumption, family behavior and habits regarding eating and exercise, moderate and vigorous physical activity, sedentary behavior, local foods and environment factors that impact the family. In addition, the child's weight will be measured at each time point.

Participation in La Vida Buena will take 6 months. At the Nogales site, participants will be invited to a series of weekly classes over the course of 8 weeks that are being offered by the Mariposa clinic related to child healthy weight, exercise and nutrition. At the Rio Rico site, participants will be offered one face to face educational session about child healthy weight with Mariposa staff. Participants will be scheduled for BMI measurements and questionnaires three months after initiating the program, as well as six months after initiating the La Vida Buena Program.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 8 years of age
* Above the 85th percentile for obesity
* Accompanied by a parent or legal guardian.

Exclusion Criteria:

* Not between the ages of 5 and 8
* Not above the 85th percentile for obesity.
* Not accompanied by a parent or legal guardian.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
BMI | baseline to 6 months follow up
  Weight and height measured at baseline, post intervention and 6 months.

SECONDARY OUTCOMES:
Physical activity | baseline to 6 months follow up
  Increased physical activity as measured by the International Physical Activity Questionnaire - Short Form
Fruit and vegetable consumption | baseline to 6 months follow up
  As measured by self reported servings per day or week with higher values considered to be a better outcome
Simple carbohydrate consumption | baseline to 6 months follow up
  As measured by self report servings per day or week with lower values considered to be a better outcome
Family healthy habits | baseline to 6 months follow up
  As measured by the Family Nutrition and Physical Activity Tool designed to capture healthy family habits. The adapted scale includes 16 items that are score from 1 to 4 that measure physical activity, sport participation, television viewing and video games for their negative influence on child hood obesity. Total score ranges from 16 to 64 points, with an increased score being associated with positive outcomes. There is not threshold or cutoff for the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Maia Ingram, Principal Investigator — University of Arizona
Locations (1):
- Mariposa Community Health Center, Nogales, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is currently no plan in place, however in the future the data dictionaries and individual participant data will be available upon request

REFERENCES:
- [Derived] Tucker KM, Ingram M, Doubleday K, Piper R, Carvajal SC. La Vida Buena (The Good Life) evaluation: a quasi experimental intervention of a community health worker-led family-based childhood obesity program for Latino children 5-8 years of age on the US-Mexico border. BMC Public Health. 2019 Jun 14;19(1):759. doi: 10.1186/s12889-019-7081-x. PMID 31200685